CLINICAL TRIAL: NCT03601611
Title: Checkpoint Inhibitor Induced Colitis and Arthritis -Immunomodulation With IL-6 Blockade and Exploration of Disease Mechanisms
Acronym: COLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Inna Chen, MD, Principal Investigator, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA 1820
Record Dates: First submitted 2018-07-01; First posted 2018-07-26 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Solid Tumor; Colitis; Arthritis
MeSH Terms: conditions — Colitis; Arthritis | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: - Patients will receive tocilizumab 8 mg/kg given as an IV infusion over 60 minutes every 4 weeks (Q4W) for at least 2 cycles or until worsening or lack of improvement of diarrhea and/or colitis and/arthritis, in case of unacceptable toxicity, withdrawal of consent or clear clinical deterioration, according to investigator's judgment.
  At the initial stage, 7 patients will be enrolled and evaluated for symptom improvement. In case of ≤ 4 patients with at least one grade improvement, accrual will be terminated. If ≥ 5 patients with at least one grade improvement will be observed at the first stage, 13 additional patients will be entered at the second stage to achieve a target sample size of 20 evaluable patients. Further exploration of the treatment strategy is warranted, if at least one grade improvement is observed for ≥14 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Tocilizumab 8 mg/kg is to be given as an IV infusion over 60 minutes every 4 weeks (Q4W).
  Interventions: Drug: Tocilizumab (RoACTEMRA®)

INTERVENTIONS:
Drug: Tocilizumab (RoACTEMRA®) — Prednisolon will be given in case of worsening of symptoms
  Other Names: Prednisolon

SUMMARY:
Immune checkpoint inhibitors (ICI) might induce inflammatory potentially serious and even lethal immune related Adverse Events (irAEs). Diarrhea and/or colitis are ones of the most frequently reported irAEs in patients taking ICI. Although the immune mechanisms underlying irAEs have not been fully elucidated, studies suggest that Th17 and Tregs cells, increases in expression of immunologically-related genes, eosinophilia, microbiome among others and cytokines may be involved in the pathophysiology of immune-related complications in some diseases that resemble irAEs, such as colitis and rheumatic manifestations. Importantly, interleukin-6 (IL-6) promotes the differentiation of naïve CD4+ T cells into Th17 cells (17), and IL-6 inhibition may rebalance the altered Th17-Treg axis without inhibiting the Th1-CD8+ T-cell subsets that govern antitumor immunity. These findings raise the possibility of using IL-6 blockade as a strategy for treating colitis and arthritis induced by immune checkpoint blockade.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICI) targeting cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) and the programmed cell death protein-1 (PD-1)/programmed cell death ligand-1 (PD-L1) pathway might induce inflammatory potentially serious and even lethal immune related Adverse Events (irAEs). Diarrhea and/or colitis are ones of the most frequently reported irAEs in patients taking ICI, occurring after an average of three infusions. The incidence is higher among patients taking combination anti-CTLA-4/ anti-PD-1 therapy (44%) than those receiving anti-CTLA-4 (23-33%) or anti-PD-1 (≤19%) monotherapy. The most common autoimmune and musculoskeletal irAEs reported in clinical trials are represented by arthralgia and arthritis. The incidence of arthralgia and/or inflammatory arthritis secondary to nivolumab therapy ranges from 5% to 16% and 5%, respectively. Although the immune mechanisms underlying irAEs have not been fully elucidated, studies suggest that Th17 and Tregs cells, increases in expression of immunologically-related genes, eosinophilia, microbiome among others and cytokines may be involved in the pathophysiology of immune-related complications in some diseases that resemble irAEs, such as colitis and rheumatic manifestations. Previous studies report Th-17, that drives interleukin-17 (IL-17) production, as a key mediator of many immune diseases, including inflammatory bowel disease and ICI-induced colitis, and IL-17 elevations have been observed in experimental colitis. Importantly, interleukin-6 (IL-6) promotes the differentiation of naïve CD4+ T cells into Th17 cells (17), and IL-6 inhibition may rebalance the altered Th17-Treg axis without inhibiting the Th1-CD8+ T-cell subsets that govern antitumor immunity. An imbalance of Th17/Treg may cause the onset and progression of immune-mediated side effects. Thus, a 3-fold increase of IL-17 and IL-6 by week 12, concomitant with the development of fulminant colitis has been reported in a patient who developed presumed ipilimumab-induced colitis. These findings raise the possibility of using IL-6 blockade as a strategy for treating colitis and arthritis induced by immune checkpoint blockade.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects must have signed and dated an IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Patients with solid tumors treated with PD-1, PD-L1 and /or CTLA-4 inhibitors
* Diarrhea and/or colitis CTCAE grade ˃ 1 and/or arthritis CTCAE grade ˃ 1 induced by PD-1, PD-L1 and /or CTLA-4 inhibitors
* Age 18 years and older
* ECOG/WHO Performance Status (PS) 0-1, PS of 2 due to ongoing irAEs is allowed
* White blood cell count (WBC) ≥ 2 x 10⁹/L and/or absolute neutrophil count (ANC) ≥ 1.0 x 10⁹/L
* Platelet count ≥ 50 x 10⁹/L
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
* ASAT/ALAT ≤ 5 x ULN

Exclusion Criteria:

* History of allergy to study drug component
* Patients should be excluded if they have a condition and/or other irAEs requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration
* Females of childbearing potential or males of reproductive potential who are not willing to use an effective method of contraception, such as oral, injected, or implanted hormonal methods of contraception, intrauterine device or intrauterine system, condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, cream, suppository, male sterilization, or true abstinence throughout study and for a minimum of 3 months after study drug therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Rate of at least one grade improvement using the NCI CTCAE v5.0 | 2 months
  Clinical benefit of IL-6 inhibition by tocilizumab on diarrhea and/or colitis and/or arthritis induced by checkpoint inhibitors in patients with solid tumors within 8 weeks of treatment start

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months
  Safety and tolerability of the treatment regimens assessed by a summary of adverse events and clinical laboratory assessments
Rate of at least one grade improvement without prednisolone using the NCI CTCAE v5.0 | 2 months
  Clinical benefit of IL-6 inhibition by tocilizumab on diarrhea and/or colitis and/or arthritis induced by checkpoint inhibitors in patients with solid tumors without corticosteroids within 8 weeks of treatment start
Rate of sustained glucocorticoid-free remission | 6 months
  Prolonged sustained glucocorticoid-free remission

OTHER OUTCOMES:
Biomarkers | 6 months
  IL-6, IL-8, IL-17, CD4+ and CD 8+ T cells, Tregs, Th17 T cells, ANA RF, anti-CCP, CRP, WBC, ANC, CD163 and a profile of 90 proteins associated with cancer and inflammation (Olink array), fecal composition of the microflora, imaging changes and inflammation changes in colon if biopsies are available.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev & Gentofte University Hospital, Denmark, Herlev, Denmark

REFERENCES:
- [Derived] Holmstroem RB, Nielsen OH, Jacobsen S, Riis LB, Theile S, Bjerrum JT, Vilmann P, Johansen JS, Boisen MK, Eefsen RHL, Marie Svane I, Nielsen DL, Chen IM. COLAR: open-label clinical study of IL-6 blockade with tocilizumab for the treatment of immune checkpoint inhibitor-induced colitis and arthritis. J Immunother Cancer. 2022 Sep;10(9):e005111. doi: 10.1136/jitc-2022-005111. PMID 36096534